CLINICAL TRIAL: NCT06489366
Title: Efficacy of Semi-rigid Ureteroscopic Laser Lithotripsy in the Treatment of Proximal Ureteral Stones: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20240173
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Urolithiasis; Proximal Ureteral Stone
Keywords: Proximal ureteral stones; Ho: YAG lithotripsy; Thulium Fiber laser (TFL) lithotripsy; Semirigid ureteroscopic lithotripsy
MeSH Terms: conditions — Urolithiasis | interventions — Lithotripsy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients and data analysts were blinded to the allocation measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ho: YAG lithotripsy (Active Comparator): Ho; YAG laser therapy device is used. The patient adopts lithotomy position. After general anesthesia, a semi-rigid ureteroscope is used to enter the bladder through the urethra to observe the ureteral opening, and then a hydrophilic guide wire is inserted into the ureter on the affected side. After the semi-rigid ureteroscope slowly enters along the hydrophilic guide wire and reaches the bottom of the stone, the laser optical fiber of the laser therapy device is inserted into the working channel of the ureteroscope so that the end of the optical fiber is exposed in the field of view of the ureteroscope. After the laser therapy device sets the lithotripsy parameters, the optical fiber is aimed at the stone for laser lithotripsy.
  Interventions: Device: Ho: YAG lithotripsy
- Thulium Fiber laser (TFL) lithotripsy (Experimental): The patient adopts lithotomy position. After general anesthesia, a semi-rigid ureteroscope is used to enter the bladder through the urethra to observe the ureteral opening, and then a hydrophilic guide wire is inserted into the ureter on the affected side. After the semi-rigid ureteroscope slowly enters along the hydrophilic guide wire and reaches the bottom of the stone, the laser fiber of the laser therapy machine is inserted into the working channel of the ureteroscope so that the end of the fiber is exposed to the field of view of the ureteroscope. Using the TFL laser therapy device, after setting the lithotripsy parameters, the fiber is aimed at the stone for laser lithotripsy.
  Interventions: Device: Thulium Fiber laser (TFL) lithotripsy

INTERVENTIONS:
Device: Thulium Fiber laser (TFL) lithotripsy — Patients with proximal ureteral stones undergoing ureteroscopic lithotripsy using thulium laser lithotripsy.
  Arms: Thulium Fiber laser (TFL) lithotripsy
Device: Ho: YAG lithotripsy — Ho:YAG laser lithotripsy was used in patients with proximal ureteral stones undergoing ureteroscopic lithotripsy.
  Arms: Ho: YAG lithotripsy

SUMMARY:
The efficacy of Ho: YAG and TFL combined with semirigid ureteroscopic treatment of proximal ureteral stones will be compared.

DETAILED DESCRIPTION:
The target population of this study is patients with proximal ureteral stones who are scheduled to undergo semirigid ureteroscopic laser lithotripsy. After enrollment, the subjects will be randomly assigned to the semirigid ureteroscopic holmium laser (Ho: YAG) lithotripsy group and the semirigid ureteroscopic thulium fiber laser (TFL) lithotripsy group for surgical treatment. The subjects will be followed up after surgery, and the collected data will be summarized and analyzed after the study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. patients diagnosed with unilateral proximal ureteral stones ≤2cm by computed tomography (CT)/Kidney and upper bladder (KUB) radiography who required surgery;
3. patients who volunteered to participate in this study.

Exclusion Criteria:

1. Unable to give informed consent;
2. Untreated urinary tract infection;
3. Pregnant women;
4. Known anatomical abnormalities (such as urinary diversion or ureteral stenosis);
5. Urothelial tumors, transplanted kidney stones, irreversible coagulopathy;
6. The semi-rigid ureteroscope cannot reach the stone site, ureteroscopy-negative stones, and stones can be removed directly without laser lithotripsy;
7. The researchers believe that they are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-06-26 (Estimated); Primary Completion 2025-01-26 (Estimated); Study Completion 2025-02-26 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate (SFR) | 2-4 weeks after surgery
  Stone-free rate (SFR) after single-session laser lithotripsy using a semirigid ureteroscope without an auxiliary procedure assessed by CT/X-ray at 2-4 weeks follow-up after laser lithotripsy.

SECONDARY OUTCOMES:
Operative time | Immediately during surgery
  the time of laser lithotripsy
Intraoperative complications | Immediately during surgery
  bleeding, ureteral perforation, ureteral wall injury, or intraoperative adverse events leading to termination of surgery
Postoperative complications | 2-4 weeks after surgery
  Occurrence of postoperative complications
Additional procedures | Intraoperatively and before removal of the Ureteral stents
  If semi-rigid ureteroscopy combined with laser lithotripsy fails, it is converted to flexible ureteroscopy, PCNL, laparoscopic lithotomy. In addition, ESWL treatment is performed before the double-J stent is removed after surgery.lithotripsy, and postoperative ESWL treatment before removal of the ureteral stents, among others.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital, Wuhan University,, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No